CLINICAL TRIAL: NCT04715815
Title: Effects of COVID-19 on Chronic Pain Patients in Terms of Pain and Pain Management
Brief Title: COVID-19 and Its Effects on Chronic Pain Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sasikaan Nimmaanrat, Primary Investigator, Head of Pain Clinic, Clinical Associate Professor, Prince of Songkla University
Other Study IDs: REC.63-359-8-1
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention (only interview) — Interview

SUMMARY:
Pain is an unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage. Many factors can affect pain and its severity.

This study aims to explore how the COVID-19 affects chronic pain patients in terms of pain in general, intensity of pain, desire for pain treatment including follow up visits and pain medication refills as well as sleep.

DETAILED DESCRIPTION:
Research question

What are the effects of the COVID-19 on chronic pain patients in terms of pain and pain management?

Conceptual framework

The COVID-19 is a novel emerging infectious disease which has unimaginable and unbelievable large scale distressing effects worldwide.

Up to date, there is no study which aims to evaluate the effects of the COVID-19 on chronic pain patients in terms of pain and pain management. The previous survey in patients focused on the worrisome of them for getting this infection and their confidence in their government to control the COVID-19 situation in the US.

Materials and methods

This study is an in-depth interview. The in-depth interview is the principal method to collect qualitative data by setting up open-ended questions beforehand. Patients who are interviewed, can express their attitudes freely. This method is flexible which words, sentences and questions can be adjusted to suit each interviewee (participant). The process consists of active and intentional listening as well as ask on an in-depth basis. All conversations during the in-depth interview are tape-recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pain who have been under the health care service of the pain clinic of Songklanagarind hospital.
* Chronic pain patients are patients with persistent pain for at least 3 months. Pain can be from any etiologies.
* The expected number of interviwees for this in-depth interview is 30 or until the gathered interview data are saturated.

Exclusion Criteria:

* Patients who are not willing to participate this study and have time for an in person 'in-depth interview'.
* Patients who are not influence in Thai language.
* Patients who are physically or mentally too ill to participate this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older who have chronic pain for at least 3 months' duration.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
To explain how the COVID-19 affects chronic pain patients in terms of pain and pain management. | January to December 2021
  An in-depth interview will be conducted to find out how the COVID-19 affects chronic pain patients. The investigators will measure pain intensity and sleep disturbance level by using an 11-point numerical rating scale where 0 means that the patient's pain condition is not affected by the COVID-19 and 10 means that the patient's pain condition is maximally affected. The higher the score is the worse.

SECONDARY OUTCOMES:
To explain how the COVID-19 affects chronic pain patients' psychological status. | January to December 2021
  An in-depth interview will be performed to find out how the COVID-19 affects the psychological aspect of chronic pain patients. The level of anxiety and stress will be measured using the 11-point verbal numerical rating scale where 0 means that the patient's psychological status is not affected by the COVID-19 and 10 means that the patient's psychological status is maximally affected. The higher the score is the worse.

CONTACTS AND LOCATIONS:
Overall Officials: Sasikaan Nimmaanrat, MD, Principal Investigator — Faculty of Medicine, Prince of Songkla University

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon request.

REFERENCES:
- [Result] Wolf MS, Serper M, Opsasnick L, O'Conor RM, Curtis L, Benavente JY, Wismer G, Batio S, Eifler M, Zheng P, Russell A, Arvanitis M, Ladner D, Kwasny M, Persell SD, Rowe T, Linder JA, Bailey SC. Awareness, Attitudes, and Actions Related to COVID-19 Among Adults With Chronic Conditions at the Onset of the U.S. Outbreak: A Cross-sectional Survey. Ann Intern Med. 2020 Jul 21;173(2):100-109. doi: 10.7326/M20-1239. Epub 2020 Apr 9. PMID 32271861